CLINICAL TRIAL: NCT06828549
Title: MObile Support Adapted to Individual Contexts (MOSAIC Study)
Brief Title: MObile Support Adapted to Individual Contexts
Acronym: MOSAIC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lindsay Mayberry, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 242066; 1R01DK140190-01 (NIH)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: family support; social support; text message; mobile health; hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Mosaicism; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The labs analyzing A1c results (primary outcome, hemoglobin A1c) are marked to the study description or participants' assigned condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MOSAIC (Experimental): PWD participants will receive MOSAIC components (monthly phone coaching and text message support for goals and medication adherence) for 12 months. PWD participants will receive high-quality print materials upon enrollment and quarterly newsletters on healthy living with diabetes.
  All SP participants invited by PWD participants assigned to MOSAIC will receive high-quality print materials upon enrollment and quarterly newsletters on healthy living with diabetes. SPs may participate in monthly phone coaching and/or receive text message support tailored to the goal set by the linked PWD.
  Interventions: Behavioral: MOSAIC; Behavioral: Print Materials
- Print Materials (Placebo Comparator): PWD participants will receive text messages advising how to access their study A1c test results, and receive high-quality print materials including a book upon enrollment and quarterly newsletters on health living with diabetes.
  Interventions: Behavioral: Print Materials

INTERVENTIONS:
Behavioral: MOSAIC — All MOSAIC PWD participants receive monthly phone coaching following a semi-structured protocol plus daily automated text message support. MOSAIC uses the mobile phone-delivered structure and functionality developed for FAMS (NCT04347291). Tailoring rules novel to MOSAIC determine phone coaching protocol content, text message content, and the involvement of a SP. Semi-structured protocols used in prior studies (and in the case of NCT04334109 adapted for mobile phone-delivery) are employed. Per tailoring rules, enrolled SPs may be invited to participate in monthly coaching calls with the PWD and/or receive text messages about supporting the PWD. The study will not assess outcomes or effects among SPs.
  Other Names: Family/friend Activation to Motivate Self-Care (FAMS; NCT04347291); Family Diabetes Self-Management Education and Support (NCT04334109); Standard Diabetes Self-Management Education and Support (NCT04334109); Diabetes Distress Reduction
  Arms: MOSAIC
Behavioral: Print Materials — Quality print materials about diabetes management provided upon enrollment and in quarterly study newsletters

SUMMARY:
This behavioral clinical trial evaluates an adaptively tailored, mobile phone-delivered intervention (MOSAIC) designed to support adults managing their type 2 diabetes. Adaptive means the intervention can change over time. Tailored means the intervention may be different for different participants. The main questions the study will aim to answer are:

1. Does the diabetes education and support delivered via the MOSAIC adaptive mobile phone-delivered intervention improve outcomes more than diabetes education and support delivered via print materials alone? This aim compares the study arms on outcomes such as glycemic management (hemoglobin A1c), diabetes distress, and psychosocial well-being. This aim also compares the study arms on intervention targets (mediators) including diabetes self-efficacy and self-care behaviors.
2. For whom does the MOSAIC adaptive tailoring approach improve outcomes more than the print materials alone? This aim examines how well the tailoring rules used for the MOSAIC intervention worked for different participants on the outcomes examined in the first aim.

Participants will enroll in a 16-month study with assessments every 4 months. Assessments include completion of an A1c test and a survey. For those assigned to MOSAIC, they will experience 12-months of mobile phone-delivered support with 3 opportunities for intervention tailoring.

DETAILED DESCRIPTION:
MOSAIC intervention components include:

* Monthly coaching sessions (~30 minutes each) - Persons with diabetes (PWD) will engage in goal setting and skill building relevant to their self-identified diet, exercise, and/or stress management goal
* Daily one-way and interactive text messages to support the PWD in meeting their goal and supporting medication adherence
* Weekly interactive text messages asking the PWD to reflect on goal progress followed by personalized feedback from their coach
* The option to invite an adult support person (SP). SPs may be invited to participate in monthly phone coaching and/or receive text messages (3 one-way texts per week and one interactive text per week) pertaining to supporting the PWD, per the MOSAIC intervention adaptive tailoring rules

PWD participants will be randomized in a parallel design to the MOSAIC adaptive mobile phone-delivered intervention or to print materials alone. The study is powered to detect a 0.5% reduction in hemoglobin A1c. Analyses will examine effects during the intervention (4 and 8 months) and post-intervention (12 months) and sustained effects (16 months). Participants will be analyzed as randomized regardless of withdrawal from the intervention (i.e., intention-to-treat principals) and missing data will be imputed.

ELIGIBILITY:
Inclusion Criteria:

PERSONS WITH DIABETES:

* Speaks and reads in English
* 18-75 years old
* Diagnosed with type 2 diabetes
* Receiving outpatient care from a partnering clinic
* Community-dwelling (e.g., not in a nursing facility)
* Prescribed at least one daily diabetes medication
* Owns a mobile phone

SUPPORT PERSONS:

* Speaks and reads in English
* 18 years or older
* Owns a mobile phone

Exclusion Criteria:

PERSONS WITH DIABETES:

* Unable to communicate by phone
* Currently pregnant
* Currently undergoing treatment for cancer (e.g., radiation, chemotherapy)
* Diagnosed with end-stage renal disease
* Receiving hospice services*
* Diagnosed with congestive heart failure
* Diagnosed with dementia
* Diagnosed with schizophrenia
* Demonstrated an inability to receive and respond to a text
* Does not take medication on his/her own/medication administered by someone else

SUPPORT PERSONS:

* Demonstrated inability to receive & respond to a text
* Unable to communicate by phone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c During Intervention Period | Baseline and 4, 8, and 12 months post-baseline
  Hemoglobin A1c assessed by mail-in A1c kits from BioQuintex and/or taken from electronic health record (venipuncture or point-of-care) where higher values indicate worse glycemic management
Change in Hemoglobin A1c Sustained Post-intervention Effects | Baseline and 16 months post-baseline
  Hemoglobin A1c assessed by mail-in A1c kits from BioQuintex and/or taken from electronic health record (venipuncture or point-of-care) where higher values indicate worse glycemic management

SECONDARY OUTCOMES:
Change in Diabetes Distress During Intervention Period | Baseline and 4, 8, and 12 months post-baseline
  Assessed by the Problem Areas in Diabetes (PAID-5) with scores ranging 0-100 where higher scores indicate more emotional, psychological and social distress related to diabetes management (worse)
Change in Diabetes Distress Sustained Post-intervention Effect | Baseline and 16 months post-baseline
  Assessed by the Problem Areas in Diabetes (PAID-5) with scores ranging 0-100 where higher scores indicate more emotional, psychological and social distress related to diabetes management (worse)
Change in Psychosocial Well-being During Intervention Period | Baseline and 4, 8, and 12 months post-baseline
  Assessed by the World Health Organization - Five Well-Being Index (WHO-5) with scores ranging 0 to 100 where higher scores indicate more well-being (better)
Change in Psychosocial Well-being Sustained Post-intervention Effect | Baseline 16 months post-baseline
  Assessed by the World Health Organization - Five Well-Being Index (WHO-5) with scores ranging 0 to 100 where higher scores indicate more well-being (better)

OTHER OUTCOMES:
Change in Diabetes Self-efficacy (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  as assessed by the Perceived Diabetes Self-Management Scale with scores ranging 8 to 40 with higher scores indicating more self-efficacy (better)
Change in Diabetes Self-care Quality (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  Diabetes Self-Management Questionnaire - Revised (DSMQ-R) with scores ranging 0-10 with higher scores indicating more effective self-care behaviors (better)
Change in Dietary Behavior (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  as assessed by Personal Diabetes Questionnaire, Use of Information for Decision Making Scale with scores ranging 1-6 where higher scores indicate more use of dietary information for decision making (better)
Change in Dietary Behavior (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  as assessed by Personal Diabetes Questionnaire, Problem Eating Behavior scale with scores ranging 1-6 where higher scores indicate more problem eating behaviors (worse)
Change in Physical Activity (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  As assessed by the Physical Activity Scale for the Elderly (PASE) with scores ranging 0-400 where higher scores reflect greater levels of physical activity (better)
Change in Physical Activity (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  As assessed by the Exercise Vital Sign (EVS) with scores ranging 0-1,050 minutes per week of moderate to strenuous physical activity where higher scores indicate more physical activity (better)
Change in Diabetes Medication Adherence (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  as assessed by the Summary of Diabetes Self-Care Activities medications subscale with scores ranging 0 to 7 representing days in the prior week with perfect adherence (higher is better)
Change in Diabetes Medication Adherence (Outcome & Mediator) | Baseline and 4, 8, 12, and 16 months post-baseline
  as assessed by the Adherence to Refills and Medications in Diabetes scale, with scores ranging 11-44 with higher scores indicating more problems with adherence (worse)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials, de-identified individual and aggregate survey, clinical, and laboratory data (including raw and recoded data) and associated study documentation (survey codebook; analytic code used in survey and clinical data analyses; standard citation and unique identifier to facilitate attribution of data use) will be made publicly available through the Open Science Framework (OSF).
Supporting Information: SAP, Analytic Code
Time Frame: After study results are posted on clinical trials (required to occur within 1 year of final data collection), scientific data will be submitted to the Open Science Framework (OSF). Under the current repository policies, data will be preserved and available for the wider research community in perpetuity.
Access Criteria: Survey, clinical, and laboratory data and associated study documentation (survey codebook; analytic code used in survey and clinical data analyses; standard citation and unique identifier to facilitate attribution of data use) will be shared and made publicly available through OSF as open access. Survey, clinical, and laboratory data will be made available in csv and text format and will not require the use of specialized tools to be accessed or manipulated. All shared data and documentation will be findable and identifiable using the standard data indexing tools in Open Science Framework.